CLINICAL TRIAL: NCT01420679
Title: A Multi-center, Randomized, Phase 3 Study of Sequential Pralatrexate Versus Observation in Patients Previously Undiagnosed Peripheral T-cell Lymphoma Who Achieved an Objective Response After Initial Treatment With CHOP-based Chemotherapy
Brief Title: Pralatrexate vs Observation Following CHOP-based Chemotherapy in Undiagnosed Peripheral T-cell Lymphoma Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDX-017; 2010-022230-81 (EudraCT Number)
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Lymphoproliferative Disorders; Lymphoma; Non-Hodgkin's Lymphoma; T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoproliferative Disorders; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell | interventions — 10-propargyl-10-deazaaminopterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pralatrexate (Experimental): Patients randomized to the Pralatrexate Arm will receive pralatrexate injection and Vitamins B12 and Folic Acid until a criterion for pralatrexate injection treatment discontinuation is met.
  Interventions: Drug: Pralatrexate Injection
- Observation (No Intervention): Patients randomized to the Observation Arm will receive Vitamins B12 and Folic Acid and remain under observation until a criterion for observation discontinuation is met.

INTERVENTIONS:
Drug: Pralatrexate Injection — Intravenous (IV) push administration over 30 seconds to 5 minutes via a patent IV line containing normal saline (0.9% sodium chloride).
  Initial dose: 30 mg/m2
  Administered weekly for 3 weeks of a 4-week cycle until criteria for discontinuation per the protocol are met.
  Other Names: FOLOTYN; PDX; Pralatrexate; (RS)-10-propargyl-10-deazaaminopterin
  Arms: Pralatrexate

SUMMARY:
The purpose of this study is to see if pralatrexate extends response and survival following CHOP-based chemotherapy (CHOP: cyclophosphamide, doxorubicin, vincristine, and prednisone) and if pralatrexate improves response in patients with partial response following CHOP-based chemotherapy. Patients will either receive pralatrexate or be under observation. All patients will receive vitamins B12 and folic acid and attend regular clinic visits to evaluate their disease and health.

DETAILED DESCRIPTION:
This was an international, multi-center, randomized, Phase 3, open-label study of sequential pralatrexate versus observation in patients with previously undiagnosed PTCL who have achieved an objective response following initial treatment with CHOP-based chemotherapy.

Upon documentation of completion of an objective response following at least 6 cycles of a designated CHOP-based chemotherapy confirmation of histopathology by independent review, and confirmation that all eligibility criteria were met, patients were randomized in a 2:1 ratio to either pralatrexate or observation, according to a permuted block design with stratification factor of Tumor Response per Investigator at completion of CHOP-based therapy (Complete Response [CR] vs Partial Response [PR]).

All patients who receive at least 1 dose of pralatrexate were followed for safety through 35 (± 5) days after their last dose of pralatrexate or until all treatment-related AEs have resolved or returned to baseline/Grade 1, whichever is longer, or until it was determined that the outcome does not change with further follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient has one of the following peripheral T-cell lymphoma (PTCL) subtypes confirmed by an independent central pathology reviewer, using the Revised European American Lymphoma World Health Organization disease classification:

  * T/natural killer (NK)-cell leukemia/lymphoma
  * Adult T-cell lymphoma (TCL)/leukemia (human T-cell leukemia virus 1+)
  * Angioimmunoblastic TCL
  * Anaplastic large cell lymphoma (ALCL), primary systemic type, excluding anaplastic lymphoma kinase positive (ALK+) with International Prognostic Index (IPI) score less than 2 at initial diagnosis and complete response (CR) after CHOP-based therapy
  * PTCL-unspecified
  * Enteropathy-type intestinal lymphoma
  * Hepatosplenic TCL
  * Subcutaneous panniculitis TCL
  * Transformed mycosis fungoides (tMF)
  * Extranodal T/NK-cell lymphoma nasal or nasal type
  * Primary cutaneous gamma-delta TCL
  * Primary cutaneous CD8+ aggressive epidermic cytotoxic TCL
* Documented completion of at least 6 cycles of CHOP-based therapy:

  * CHOP 21
  * CHOP 14
  * CHOP + etoposide
  * Other CHOP variants: substitution allowed for 1 component with a drug of the same mechanism of action. Additional components, except alemtuzumab, are allowed. Rituximab may be added if not given within 3 cycles of randomization.
* Patient has achieved CR or partial response (PR) per per investigator's assessment following completion of CHOP-based therapy and has had radiological assessment within 21 days prior to randomization.
* Eastern Cooperative Oncology Group performance status less than or equal to 2.
* Adequate blood, liver, and kidney function as defined by laboratory tests.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to randomization and agree to practice a medically acceptable contraceptive regimen from study treatment initiation until at least 30 days after the last administration of pralatrexate.
* Men who are sexually active, including those with a pregnant partner, must agree to practice a medically acceptable barrier method contraceptive regimen (eg, condoms) while receiving pralatrexate and for 90 days after the last administration of pralatrexate.
* Has given written informed consent.

Exclusion Criteria:

* Patient has:

  * Precursor T/NK neoplasms
  * ALCL (ALK+) with IPI score less than 2 at initial diagnosis and CR after CHOP-based therapy
  * T cell prolymphocytic leukemia
  * T cell large granular lymphocytic leukemia
  * Mycosis fungoides, except tMF
  * Sézary syndrome
  * Primary cutaneous CD30+ disorders: ALCL and lymphomatoid papulosis
* If there is a history of prior malignancies other than those below, must be disease free for at least 5 years. Patients with malignancies listed below less than 5 years before study entry may be enrolled if they have received treatment resulting in complete resolution of the cancer and have no clinical, radiologic, or laboratory evidence of active/recurrent disease.

  * non-melanoma skin cancer
  * carcinoma in situ of the cervix
  * localized prostate cancer
  * localized thyroid cancer
* Receipt of prior chemotherapy (CT) or radiation therapy (RT) for PTCL, other than a single allowed CHOP regimen, except:

  * Patients with nasal NK lymphoma who received local RT less than 4 weeks prior to randomization.
  * Patients with tMF who received 1 systemic single-agent CT (except methotrexate) prior to transformation.
* Prior exposure to pralatrexate.
* Receipt of systemic corticosteroids within 3 weeks of study treatment, unless patient has been taking a continuous dose of 10 mg/day or less of oral prednisone or equivalent for at least 4 weeks or as part of a CHOP prednisone taper.
* Planned use of any treatment for PTCL during the course of the study.
* Patient has:

  * Human immunodeficiency virus (HIV)-positive diagnosis with a CD4 count of less than 100 mm3 or detectable viral load within past 3 months and receiving anti-retroviral therapy.
  * Hepatitis B (HBV)-positive serology and is receiving interferon therapy or has liver function test results outside the parameters of study inclusion criteria. Other antiviral therapies are permitted if at a stable dose for at least 4 weeks.
  * Hepatitis C (HCV) virus with detectable viral load or immunological evidence of chronic active disease or receiving/requiring antiviral therapy.
  * Symptomatic central nervous system metastases or lesions requiring treatment.
  * Uncontrolled hypertension or congestive heart failure Class III/IV per the New York Heart Association's Heart Failure Guidelines
  * Active uncontrolled infection, underlying medical condition including unstable cardiac disease, or other serious illness impairing the ability of the patient to receive protocol treatment.
* Major surgery within 2 weeks prior to study entry, except for line placement or biopsy procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (3):
  - Detroit Clinical Research Center, PC, Novi, Michigan
  - New York Presbyterian Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Australia (8):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Center, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - Saint Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Cabrini Health, Malvern, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (2):
  - AZ Sint-Jan, Bruges
  - Universitair Ziekenhuis Gent, Ghent
- Canada (2):
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
- France (2):
  - Hôpital Morvan, Brest
  - CHU Haut-Leveque, Pessac
- St James Hospital, Dublin, Ireland
- Israel (4):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein-Kerem Medical Centre, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (6):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli
  - Az. Ospedaliera Universitaria S. Orsola Malpighi, Bologna
  - Spedali Civili di Brescia, Brescia
  - Ospedale S. Maria delle Croci, Ravenna
  - Università Cattolica del Sacro Cuore, Roma
  - Az. Ospedaliera Università Senese, Siena
- New Zealand (4):
  - Middlemore Hospital, Otahuhu, Auckland
  - Auckland City Hospital / Auckland University, Auckland
  - Christchurch Hospital, Christchurch
  - North Shore Hospital, Milford
- Poland (3):
  - Klinika Nowotworów Ukladu Chlonnego Centrum Onkologii Instytut Marii Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Dept of Hematology and Transplantology, Gdansk
  - Małopolskie Centrum Medyczne, Krakow
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- Spain (8):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Servicio de Hematologia, Pamplona, Navarre
  - Complejo Hospitalario Universitario A Coruña- Hospital A Coruña, A Coruña
  - Hospital General Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital de Madrid Norte-Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
- United Kingdom (11):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Poole Hospital NHS Foundation Trust, Poole General Hospital, Poole, Dorset
  - Derriford Hospital, Plymouth, England
  - Sandwell & West Birmingham Hospitals NHS Trust, West Bromwich, England
  - Antrim Area Hospital, Antrim, Northern Ireland
  - NHS Greater Glasgow and Clyde Western Infirmary, Glasgow, Scotland
  - Belfast City Hospital, Belfast
  - Velindre Hospital, Cardiff
  - Royal Liverpool University Hospital, Liverpool
  - Mount Vernon Cancer Centre, Middlesex
  - UHCW (University Hospital Coventry and Warwickshire), Warwick

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 21 participants with peripheral T-cell lymphoma (PTCL) were randomized in 2:1 ratio to Pralatrexate arm or Observation arm.
Groups:
- Pralatrexate Arm: Participants randomized to Pralatrexate Arm received pralatrexate as an intravenous (IV) push administered over a minimum of 30 seconds up to a maximum of 5 minutes via a patent free-flowing IV line containing normal saline (0.9% sodium chloride [NaCl]) weekly for 3 weeks of a 4-week cycle. Initial dose of pralatrexate was 30 milligram per meter square (mg/m^2), could be reduced to 20 mg/m^2 with potential further reductions to 15 and 10 mg/m^2 based on toxicity, along with vitamin B12, 1 milligram (mg) intramuscular (IM), every 8-10 weeks and folic acid 1-1.25 mg by mouth (po) once a day (qd) until a criterion for study treatment discontinuation was met or up to a maximum of 2 years.
- Observation Arm: Participants randomized to Observation Arm received vitamin B12, 1 mg, IM every 8-10 weeks and folic acid 1-1.25 mg by mouth qd remained under observation, by attending clinic visits every 4 weeks, and being contacted by a healthcare professional during week 2 of every 4-week period until a criterion for study treatment discontinuation was met.
Period: Overall Study
Arm/Group | Pralatrexate Arm | Observation Arm
Started | 14 | 7
Completed | 0 | 0
Not Completed | 14 | 7
Not completed — Disease Progression | 3 | 2
Not completed — Adverse Event | 4 | 0
Not completed — More Than 28 Days Between Doses of Drug | 1 | 0
Not completed — Patient Decision | 1 | 0
Not completed — Investigator Decision | 1 | 2
Not completed — Sponsor Decision | 3 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pralatrexate Arm | Observation Arm | Total
Number analyzed (Participants) | 14 | 7 | 21
Age, Continuous [Median (Full Range); unit: years] | 72.0 [51 to 83] | 61.0 [44 to 83] | 68.0 [44 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 2
  Black | 1 | 1 | 2
  Arabic | 0 | 1 | 1
  White | 10 | 5 | 15
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time in days from randomization to the date of objective documentation of progressive disease (PD) or death, regardless of cause (date of PD or death - date of randomization + 1). PFS was to be assessed according to the International Workshop Criteria (IWC) without including positron emission tomography (PET). PD was defined as any new lesion or increase by greater than or equal to (>=) 50 percent (%) of previously involved sites from nadir. Participants who were alive without a disease response assessment of PD was to be censored at their last disease assessment date or the date of randomization, whichever was later. Date of progression was not to be imputed for participants with missing tumor assessments before an assessment of PD. Participants who withdraw from treatment prior to PD were to be followed for disease status whenever possible. Participants who have no response assessments after baseline were to be censored at randomization.
Time Frame: From randomization to the date of progression of disease or death due to any cause (up to 76 months)
Population: Data for this outcome measure was not collected and analyzed due to the early termination of the study.
Arm/Group | Pralatrexate Arm | Observation Arm
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time in days from randomization to the date of death, regardless of cause (date of death - date of randomization + 1).
Time Frame: From randomization until death (up to 76 months)
Population: ITT population included all randomized participants classified according to the treatment arms into which they were randomized, regardless of the actual study treatment received (or not received).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pralatrexate Arm | Observation Arm
Number analyzed (Participants) | 14 | 7
months | NA [NA to NA] — Median and 95% CI were not estimable due to low number of participants with events. | NA [NA to NA] — Median and 95% CI were not estimable due to low number of participants with events.

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as percentage of participants with an objective response of complete response (CR) or partial response (PR), relative to disease status at the time of study entry. The percentage was to be calculated by dividing number of participants within each category of response by the number of participants with measurable disease at baseline. Objective response was assessed according to the IWC without including PET. CR was defined as complete disappearance all detectable clinical evidence of disease and disease-related symptoms if present before therapy. PR was defined as regression of measurable disease and no new sites.
Time Frame: Up to 2 years
Population: Data for this outcome measure was not collected and analyzed due to early termination of the study.
Arm/Group | Pralatrexate Arm | Observation Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Worst Grade Adverse Events (AEs), Deaths, Serious Adverse Events (SAEs), and SAEs Leading to Discontinuation of Study Treatment, and Worst Grade Laboratory Abnormalities
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. AE included both serious and non- SAEs. An AE of "Hematology and Chemistry" was collected and graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03, where Grade 3 refers to severe or medically significant but not immediately life threatening and Grade 4 refers to life-threatening consequences.
Time Frame: From first dose of study drug to 35 (±5) days after last dose of study drug for the Pralatrexate Arm, and until 35 (± 5) days after the study treatment discontinuation for the Observation Arm (Up to 2 years)
Population: Safety population included all randomized participants classified according to the actual study treatment received, regardless of random assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pralatrexate Arm | Observation Arm
Number analyzed (Participants) | 14 | 7
Participants
  Participants with Any Treatment Emergent AEs | 14 | 6
  Participants with Any Grade 3 - 4 AEs | 8 | 2
  Participants with Treatment Emergent AEs Resulting in Deaths | 1 | 0
  Participants with Treatment Emergent SAEs | 4 | 0
  Participants with Any SAEs Leading to Drug Discontinuation | 2 | 0
  Hematology:Higher Than Grade 3/4 Lab Abnormalities | 3 | 1
  Chemistry:Higher Than Grade 3/4 Lab Abnormalities | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 35 (±5) days after last dose of study drug for the Pralatrexate Arm, and until 35 (± 5) days after the study treatment discontinuation for the Observation Arm (Up to 2 years)
Description: Safety population included all randomized participants classified according to the actual study treatment received, regardless of random assignment.
Arm/Group | Pralatrexate Arm | Observation Arm
All-Cause Mortality (participants affected / at risk) | 3/14 | 1/7
Serious Adverse Events (participants affected / at risk) | 4/14 | 0/7
Other Adverse Events (participants affected / at risk) | 14/14 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pralatrexate Arm (N=14) | Observation Arm (N=7)
Cardiac arrest (Cardiac disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pralatrexate Arm (N=14) | Observation Arm (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 1
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 6 | 2
Local swelling (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 4 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Bronchitis Viral (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Viral infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Gammaglutamyltransferase increased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hypokinesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 0
Melanosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Endodontic procedure (Surgical and medical procedures) | 0 | 1
Stent removal (Surgical and medical procedures) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ichthyosis (Congenital, familial and genetic disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Decreased appetite/Anorexia (Metabolism and nutrition disorders) | 0 | 1
Mucosal inflammation/Intermittant Mucositis of Mouth (General disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to business reasons. There were no safety concerns that led to study closure. No efficacy assessments and analysis was conducted. A full statistical analysis and report were not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-10-31): https://cdn.clinicaltrials.gov/large-docs/79/NCT01420679/Prot_000.pdf
  • Statistical Analysis Plan (2012-04-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT01420679/SAP_001.pdf